CLINICAL TRIAL: NCT04122105
Title: PDE5i Use in Renal Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: iss
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Nguan, associate professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (H19-02487)
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Renal Transplant Failure
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): sildenafil administration perioperative to renal transplant
  Interventions: Drug: Sildenafil
- control (Active Comparator): renal transplant recipients
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — The intervention group will receive standard care in all capacities with the exception of sildenafil administration. The first dose (50mg) will be given 1-hour prior to the surgery. Patients will be given Sildenafil twice daily up to 3 days post-transplant.

SUMMARY:
Ischemia-reperfusion (IRI) injuries are common in renal transplantation and cause poor patient outcomes. Ischemia occurs after the donor's death and reperfusion occurs after kidney implantation. The donor kidney undergoes warm ischemia (WIT) after blood circulation stops and cold ischemia (CIT) when subjected to cold storage during transportation. Decreased blood flow leads to waste product accumulation and cellular damage. During reperfusion, reactive oxygen radicals and inflammatory processes further damage the kidney. PDE5 inhibitors increase renal blood flow and could protect the kidney during transplantation. Our study assesses the utility of giving these drugs perioperatively to reduce the effects of IRI injury.

DETAILED DESCRIPTION:
1. Purpose Renal ischemia-reperfusion injuries (IRI) are the result of multifactorial mechanisms. During ischemia, the kidney is subject to reduced blood flow, oxygen delivery, and nutrients. This leads to the accumulation of nitrogenous waste products (i.e. creatinine and blood urea nitrogen) that can lead to cellular damage, depending on the extent and duration of the ischemia. Moreover, when the kidney is reperfused there is additional damage caused by reactive oxygen radicals and inflammatory processes.

   IRI is a common feature in the presentation of a diverse range of presentations: trauma, shock, sepsis, renal transplantation, cardiovascular surgery, partial nephrectomy, and other urologic complications. Moreover, IRI of the kidney specifically can lead to acute kidney injury (AKI), acute renal failure (ARF), and subsequent chronic renal failure. In the context of renal transplantation, IRI is associated with primary nonfunction, delayed graft failure, increased acute rejection, and allograft dysfunction. It has been postulated that interventions designed at increasing vasodilation during early reperfusion could reduce the effects of IRI through improving blood flow to the transplanted kidney.

   Phosphodiesterase-5 (PDE5) inhibitors, like sildenafil citrate (Viagra) and tadalafil, are drugs generally used to treat erectile dysfunction (ED) and pulmonary hypertension. These drugs prevent the breakdown of nitric oxide (NO) by increasing levels of cyclic guanosine monophosphate (cGMP). Besides causing smooth muscle relaxation and systemic vasodilation, NO and cGMP are both believed to help reduce the extent of IRI. NO has protective vasodilatory effects; while cGMP is an important mediator in the body that causes neutrophil degranulation, inhibits platelet aggregation, regulates intracellular calcium levels, and opens mitochondrial K+ATP channels.

   A number of different studies have been undertaken that support the use of PDE5 inhibitors as a pretreatment to prevent IRI in kidneys. In particular, sildenafil's antioxidant, anti-inflammatory, and antiapoptotic properties have been shown to be renoprotective in some renal injury models. However, the majority of literature is based from animal studies; there is very little information about the clinical use of PDE5 inhibitors during human kidney transplantation. Previous studies have proven that these drugs are safe for impotent males with significant comorbidities, including those on dialysis and those who underwent kidney transplants (>6 months post-op). They have also proven that sildenafil does not affect immunosuppressive drugs (i.e. tacrolimus and cyclosporine), despite these drugs sharing a common elimination pathway; Tacrolimus' pharmacokinetics, trough levels, and half-life are not significantly changed when administered with sildenafil. However, tacrolimus does change the pharmacokinetics (increase in Cmax and half-life) of sildenafil when both are administered together.

   These studies prove that PDE5 inhibitors are renoprotective, generally well-tolerated, and do not impact immunosuppressants. However, what they have not shown is the effect of PDE5 inhibitors administered early in human kidney transplantation and their effect on the transplanted kidney. Our study will try to amend this by looking at utility of perioperative administration of sildenafil in early effects on the transplanted allograft.
2. Hypothesis A.) PDE5 inhibitors given perioperatively will decrease ischemia reperfusion injury and lead to consequently improved function in the transplanted kidney.
3. Justification In 2018, 133 transplants were performed by the Vancouver General Hospital (VGH) Kidney Transplant program. 38 of these kidneys were from living donors (LD), while the remaining 95 were cadaveric donations. This data supports that the majority of renal transplants are done using kidneys from deceased donors (DD) as opposed to LDs. However, the quality of these donated organs can vary drastically and DD organs are more likely to have poorer outcomes relative to LD. This is because the DD kidney undergoes warm ischemia (WIT) after the blood circulation is stopped and then cold ischemia (CIT) when subjected to hypothermic conditions meant to preserve the organ. The combined effects of WIT and CIT inflict cellular damage and may impair renal blood flow to cause primary renal dysfunction, delayed graft failure, increased acute rejection, and allograft dysfunction. Increased renal perfusion in this critical phase through vasodilation may counteract some of these negative effects of procurement and implantation

   There is a lot of heterogeneity among DD kidneys due to the exact cause of the donor's death. Donation after circulatory death (DCD), as opposed to donation after brain death (DBD), kidney transplants have a higher chance of delayed graft function (DGF). DGF is defined as needing dialysis in the first week of transplant. This is common in marginal donor organs such as DCD or extended criteria (ECD) cadaveric transplants and can predispose to slow graft function or delayed graft function, which themselves are associated with increased rates of acute rejection and poorer outcomes. Our study aims to look at both DCD and DBD transplants to determine if PDE5 inhibitors can positively impact graft function of DD kidneys.
4. Objective A) To measure the utility of perioperative administration of PDE5 inhibitors in kidney transplant recipients (RTRs)
5. Research Design DRUG CHOICE Sildenafil has the longest safety record of the PDE5 inhibitors. Moreover, it is shown to have a more potent effect in IRI studies. A dose of 50mg twice a day is the standard dose given to patients with Erectile Dysfunction (ED).

   METHOD A patient who has given written informed consent will be given a randomly generated subject ID that is not derived from any aspect of their personally identifying information, nor details regarding their operation. This subject ID will be stored on a master list alongside their personal health number to serve as a unique method of identifying patients.

   Patients will randomly be assigned to either the control (no PDE5 inhibitor) or the intervention (sildenafil) group. The control group will receive standard care. The intervention group will receive standard care in all capacities with the exception of sildenafil administration. The first dose (50mg) will be given 1-hour prior to the surgery. Patients will be given Sildenafil twice daily up to 3 days post-transplant.

   Data will be collected and stored on an encrypted, office-only hard drive. Information on demographics (gender, ethnicity, age, etc.) and postoperative results (kidney function, all cause 90-day perioperative morbidity and mortality, postoperative complications, and length of stay in hospital) will be recorded for all patients on an password protected Excel file.

   OUTCOMES Outcomes including intraoperative, postoperative and 90 day followup will be assessed. Intraoperative: xxxx, xxxx, xxx, xxx. Postoperative: kidney function, all cause 90-day perioperative outcomes including xxxx, xxx, xxx, xxx. Time zero biopsies are done as routine and will likewise be taken into account. Kidney Function will be determined through daily bloodwork while an inpatient, and twice a week for the first 4 weeks, once a week from weeks 5-8, and then every 2 weeks from weeks 9-12. This is the standard of care follow-up in the Program. All information is normally collected for transplant patients on this schedule and no extra time or discomfort will be required on the part of the patient.
6. Statistical Analysis This study will use the Chi square method to analyze categorical data and the t-test between groups to analyze continuous variable. A P-value < 0.05 will be considered statistically significant.

For this study, he investigators propose n=100 with 50/50 split between patients undergoing DCD and DBD transplants and a 1:1 split in the control and experimental arms. Therefore, there will be 25 patients in each of the following arms: DCD experimental, DCD control, DBD experimental, and DBD control. The VGH Kidney transplant program completed 133 transplants in 2018. Out of this, 95 were cadaveric transplants. Assuming similar numbers in the future with 50% of the recipients participating, it will take about 2 years to accrue the data needed for adequate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant patients at VGH undergoing donation after circulatory death (DCD) and donation after brain death (DBD) kidney transplants
* 19 years of age
* able to provide consent.

Exclusion Criteria:

* Patients that are unable to understand the purpose of the study or cannot give written consent will be excluded.
* Moreover, patients with contraindications to PDE5 inhibitors will be excluded from the study. PDE5 inhibitors are generally well tolerated, even in patients with severe renal disease, those on dialysis, and in transplant recipients. Patients will be excluded if they are taking nitrates of any form (contraindication), are allergic to sildenafil or any of the ingredients of this medication, are on an alpha-adrenergic blocker (potential risk)
* patients currently on any experimental drug in the last 3 months (confounding factor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
renal transplant function within 90 days postop | 90 days postop
  renal functional improvement

SECONDARY OUTCOMES:
perioperative safety of sildenafil administration in renal transplantation | intraoperative and 90 days postop
  perioperative safety of sildenafil administration to renal transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No